CLINICAL TRIAL: NCT00280722
Title: Does Increasing Research Awareness Impact on Accrual? A Feasibility Study. Protocol Version 3.4 Dated April 2005.
Brief Title: RAW Study Version 3.4
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: Liverpool John Moores University (Other); National Cancer Research Network (Network)
Allocation: Randomized | Purpose: Other
Other Study IDs: 4858
Record Dates: First submitted 2006-01-20; First posted 2006-01-23 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2006-01

CONDITIONS: Cancer
Keywords: Randomised; Intervention; Leaflet; Information; Awareness; Behaviour; Research
MeSH Terms: conditions — Neoplasms; Behavior

INTERVENTIONS:
Behavioral: patient information leaflet

SUMMARY:
The purpose of this study is to investigate the feasibility of carrying out a full scale randomised controlled trial to compare the effects of giving additional information versus no additional information to patients prior to their first oncology appointment.

Hypothesis: Patients with some awareness of research provided prior to clinic appointment in oncology and aware of the possibility of being invited to take part in a clinical trial are more likely to agree to participate.

DETAILED DESCRIPTION:
The recruitment of cancer patients into clinical trials may be hindered by several factors such as limited understanding of medical research, a lack of information about the type of research on offer for patients, over load of information when given a new and life limiting diagnosis. Nor does the Churchill Hospital inform patients that research is an integral part of the every day life and business of the hospital.

Does increasing research awareness impact on accrual?

This initial study aims to establish the feasibility of a larger study to gather the evidence required to investigate whether patients need some information indicating that a hospital participates in research, and what it may mean to the individuals to participate, including new terminology; thus reducing fear and anxiety and ultimately increasing the accrual of cancer patients into cancer clinical trials. Prior knowledge of patients' attitudes to involvement in clinical trials might assist communication about trials and encourage more doctors to approach eligible patients. In the NHS there is always a fear of cost implications, however a study comparing two New Patient Information Packs (NPIPs) showed no differences were detected between a full pack and a mini pack and given the cost, the mini-New Patient Information Pack (mini-NPIP) was the preferred approach. This has influenced the decision to provide only a brief leaflet of information to patients prior to their first appointment.

The National Cancer Research Network (NCRN) was formed three years ago with the aim to provide the NHS infrastructure to support and improve patient care by speeding up access to the best treatment and care, provide information and support to our patients and improve the speed of research by increasing the number of patients into clinical trials. In the Thames Valley Cancer Research Network (TVCRN) accrual has increased from 2.7% in 2001-2 to 8.3% in 2003-4. The infrastructure to support research is in place, clinicians are informed and have relevant nursing and administrative support to offer trials to patients and cope with the increased numbers of patients taking part. There appears to be a deficit in the research knowledge and understanding of the general public. It is easier and less stressful to 'opt out' when faced with a new diagnosis and complicated treatment options than to consider, in addition, a clinical trial. By measuring accrual and evaluating the patients' response to information about research I intend to investigate the feasibility of a larger study to provide the evidence to investigate the need for pre-first-visit research information. Thus investigating the requirement, importance and need for information for the patients before their first oncology appointment and the general public.

Ellis, Buttow and Tattersall have published two studies conducted with breast cancer patients: the first in 2001 found that that women who have a better knowledge of clinical trials are more willing to consider participating in a clinical trial, however in 2002 patients who had received a booklet of information about research for patients were significantly less likely to consider participating in a randomised clinical trial (RCT). Using a very large sample (n=2331) Jenkins, Fallowfield and Saul showed that the vast majority of cancer patients questioned wanted a great deal of specific information concerning their illness and treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient requiring first oncology appointment whose appointments are being planned more than 3 days in advance. (see exclusion criteria for reason)
2. 18 years or over. (The project will take place in adult clinic - all children & young people under 18 are seen and cared for in the paediatric unit.) -

Exclusion Criteria:

1. New patient referrals whose appointments are being planned in less than 3 days are often telephoned with details and will not have sufficient time to receive the information by post and read it prior to their appointment.
2. Vulnerable patients under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-01; Study Completion 2006-11 (Estimated)

PRIMARY OUTCOMES:
Whether it is feasible to carry out a full scale randomised controlled trial to compare the effect of giving additional information versus no additional information to patients prior to their first oncology appointment.

SECONDARY OUTCOMES:
Whether existing and/or acquired research awareness may influence participation.
Development of the research information leaflet.
Development, testing and validation of the data collection methods.
Number of questionnaires returned.
Realistic data for estimating sample sizes in the larger study.

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Palmer, Principal Investigator — Thames Valley Cancer Research Network
Locations (1):
- Churchill Hospital, Oxford, United Kingdom

REFERENCES:
- [Background] Stevens T, Ahmedzai SH. Why do breast cancer patients decline entry into randomised trials and how do they feel about their decision later: a prospective, longitudinal, in-depth interview study. Patient Educ Couns. 2004 Mar;52(3):341-8. doi: 10.1016/S0738-3991(03)00041-7. PMID 14998605
- [Background] Fallowfield LJ, Jenkins V, Brennan C, Sawtell M, Moynihan C, Souhami RL. Attitudes of patients to randomised clinical trials of cancer therapy. Eur J Cancer. 1998 Sep;34(10):1554-9. doi: 10.1016/s0959-8049(98)00193-2. PMID 9893627
- [Background] Mohide EA, Whelan TJ, Rath D, Gafni A, Willan AR, Czukar D, Campbell IB, Okawara GS, Neimanis M, Levine MN. A randomised trial of two information packages distributed to new cancer patients before their initial appointment at a regional cancer centre. Br J Cancer. 1996 Jun;73(12):1588-93. doi: 10.1038/bjc.1996.299. PMID 8664135
- [Background] Ellis PM, Butow PN, Tattersall MH, Dunn SM, Houssami N. Randomized clinical trials in oncology: understanding and attitudes predict willingness to participate. J Clin Oncol. 2001 Aug 1;19(15):3554-61. doi: 10.1200/JCO.2001.19.15.3554. PMID 11481363
- [Background] Ellis PM, Butow PN, Tattersall MH. Informing breast cancer patients about clinical trials: a randomized clinical trial of an educational booklet. Ann Oncol. 2002 Sep;13(9):1414-23. doi: 10.1093/annonc/mdf255. PMID 12196367
- [Background] Jenkins V, Fallowfield L, Saul J. Information needs of patients with cancer: results from a large study in UK cancer centres. Br J Cancer. 2001 Jan 5;84(1):48-51. doi: 10.1054/bjoc.2000.1573. PMID 11139312
- [Background] Harrison J. Why it is preferable to learn before the moment of diagnosis. In: Marie Curie Cancer Care in association with the Consumers' Advisory Group for Clinical Trials (CAG-CT) Conference: Towards Public Understanding of Clinical Trials, 16 Feb 1998, London.
- [Background] Blesing C, Palmer S, Mathews A. Thames Valley Cancer Research Network 3rd Annual Progress Report. 2004. http://www.tvcn.org.uk/research/annualreport.
- [Background] Mossman J, Boudioni M, Slevin ML. Cancer information: a cost-effective intervention. Eur J Cancer. 1999 Oct;35(11):1587-91. doi: 10.1016/s0959-8049(99)00195-1. PMID 10673966
- [Background] Braunholtz DA, Edwards SJ, Lilford RJ. Are randomized clinical trials good for us (in the short term)? Evidence for a "trial effect". J Clin Epidemiol. 2001 Mar;54(3):217-24. doi: 10.1016/s0895-4356(00)00305-x. PMID 11223318